CLINICAL TRIAL: NCT05042635
Title: A Multi-center, Randomized, Double-blind Controlled Study on the Sequential Treatment of Psoriasis With Traditional Chinese and Western Medicine
Brief Title: Sequential Treatment of Psoriasis With Traditional Chinese and Western Medicine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Collaborators: Shanghai Skin Disease and Venereal Disease Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21Y21920100
Record Dates: First submitted 2021-09-04; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Plaque Psoriasis
Keywords: Plaque Psoriasis; Ixekizumab; Jueyin granules; Randomized controlled trial; Traditional Chinese medicine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ixekizumab (4 weeks) + Jueyin Granules (12 weeks) (Experimental): Subjects received Ixekizumab in the first 4 weeks (biologic treatment period); After the cessation of biologic treatment, only Jueyin Granules was used in the 12-week traditional Chinese medicine treatment period.
  Interventions: Drug: Ixekizumab+Jueyin Granules
- Ixekizumab (4 weeks) + Jueyin placebo Granules(12 weeks) (Placebo Comparator): Subjects received Ixekizumab in the first 4 weeks (biologic treatment period); After the cessation of biologic treatment, only Jueyin placebo Granules was used in the 12-week traditional Chinese medicine treatment period.
  Interventions: Drug: Ixekizumab+Jueyin placebo Granules

INTERVENTIONS:
Drug: Ixekizumab+Jueyin Granules — Ixekizumab：160mg was injected subcutaneously at week 0 (80mg twice), then 80mg at week 2 and 4 (once).
  Jueyin Granules：Put each bag of daily dose into the same container, pour about 50ml warm water into it, stir until the particles are basically dissolved, then add proper amount of boiling water to dilute it, take it warm in two times.
  Arms: Ixekizumab (4 weeks) + Jueyin Granules (12 weeks)
Drug: Ixekizumab+Jueyin placebo Granules — Ixekizumab：160mg was injected subcutaneously at week 0 (80mg twice), then 80mg at week 2 and 4 (once).
  Jueyin placebo Granules：Put each bag of daily dose into the same container, pour about 50ml warm water into it, stir until the particles are basically dissolved, then add proper amount of boiling water to dilute it, take it warm in two times.
  Arms: Ixekizumab (4 weeks) + Jueyin placebo Granules(12 weeks)

SUMMARY:
The purpose of this study is to objectively and standardly evaluate the clinical efficacy and safety of sequential treatment of psoriasis with traditional Chinese and Western medicine through a multi-center, randomized, double-blind, placebo-controlled trial.

DETAILED DESCRIPTION:
Psoriasis is a chronic, recurrent, inflammatory disease. The incidence of this disease is increasing year by year, seriously affecting people's quality of life. Biologic agents have the advantages of rapid and efficient treatment of moderate and severe psoriasis, but their safety and recurrence are still seriously affect the application. Traditional Chinese medicine treatment of psoriasis has the advantages of fewer adverse reactions, low recurrence rate and improvement of patients' systemic symptoms while exerting the curative effect. The prevention and treatment of psoriasis by combining traditional Chinese and Western medicine has become the academic consensus. The sequential treatment of psoriasis with biological agents combined with Traditional Chinese medicine has a better therapeutic effect than that of single therapy. At present, the sequential treatment of psoriasis with targeted biological agents combined with traditional Chinese medicine has not been reported in the literature, and there is a lack of high-level clinical evidence to support it. Therefore, this project aims to provide evidence support for the clinical efficacy and safety of sequential treatment of psoriasis by traditional Chinese and Western medicine through a multi-center, randomized, double-blind, placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. It conforms to the western diagnostic criteria of plaque psoriasis and the diagnostic criteria of TCM syndrome of blood heat syndrome;
2. Physician global assessment (PGA) ≥3, psoriasis area and severity index (PASI) score ≥12, and body surface area (BSA) ≥ 10% at screening and baseline;
3. Aged between 18 and 70;
4. Those who voluntarily participate in the study and sign the informed consent.

Exclusion Criteria:

1. Erythrodermic psoriasis patients, arthropathic psoriasis patients, pustular psoriasis patients;
2. There are other active skin diseases that may affect the evaluator;
3. Have systematically received other investigational drugs within 1 month;
4. Received external glucocorticoid and phototherapy within 2 weeks;
5. During a period of severe and uncontrollable local or systemic acute or chronic infection;
6. Infected persons with tuberculosis;
7. Patients with viral hepatitis;
8. Serious systemic disease; Or clinical test indicators belong to one of the following cases of patients: alanine aminotransferase or glutamic-oxalacetic transaminase increase > 1.5 times the upper limit of normal value; Creatinine increase > 1.5 times the upper limit of normal value; Any one of the major blood routine indicators (white blood cell count, red blood cell count, hemoglobin amount, platelet count) is lower than the lower limit of normal value; Or other abnormal laboratory tests determined by the investigator to be unsuitable for the study;
9. Patients with a history of malignant tumor and patients with primary or secondary immune deficiency and hypersensitivity;
10. Participants in clinical trials of other drugs within 3 months;
11. Those who have undergone major surgery within 8 weeks or will require such surgery during the study period;
12. For fertile women of childbearing age who did not use highly effective contraception from the screening period until the end of the last dose;
13. Pregnant or lactating women;
14. Persons with a history of alcohol, drug or substance abuse;
15. Persons with a serious history of mental illness or family history;
16. For other reasons, the researcher considers it inappropriate to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Psoriasis area and severity index (PASI) | Up to 168 days after treatment
  Psoriasis area and severity index (PASI) score and recurrence assessment. Psoriasis area and severity index (PASI) scores were assessed for all patients at each follow-up. Recurrence was defined as a 50% reduction in maximum PASI improvement from baseline at week 40.

SECONDARY OUTCOMES:
Body surface area (BSA) | Up to 168 days after treatment
  The percentage of BSA involved in psoriasis is estimated by fingerprinting, where the entire palm of the patient represents approximately 1% of the total BSA. The number of handprints on psoriasis skin in a body part is used to determine the extent to which the body part is affected by psoriasis (%).
Physician Global Assessment (PGA) | Up to 168 days after treatment
  Physician Global Assessment (PGA)is scored on a 5-point scale, reflecting a global consideration of the erythema (E), infiltration (I),desquamation (D) across all psoriatic lesions. lt is calculated as follows: PGA score = (E +I+D) / 3 then the score needs to be rounded to the nearest whole number [PGA scale: Clear (0)-Very Severe (5)].
Dermatology Life quality index(DLQI) | Up to 168 days after treatment
  The Dermatology Life Quality Index (DLQI) is a participant-reported questionnaire used to measure the health-related quality of life (QOL) of adults suffering from a skin disease. Scores range from 0-30, a higher score indicating a greater impact on a participant's quality of life.
Patient-reported quality of life (PRQoL) | Up to 168 days after treatment
  PRQoL is used to assess the impact of psoriasis on individual social life. Scores range from 0-25, a higher score indicating a greater impact on a participant's social life.
Visual Analogue Score (VAS) | Up to 168 days after treatment
  Visual Analog Scale (VAS) is used to measure lesion pruritus from 0 to 100 mm at eash visit (with 0 being no pruritis and 100 being maximum pruritis).
CM symptom score | Up to 168 days after treatment
  The CM symptom score is used to assess changes in blood syndrome related symptoms during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Li, Study Chair — Shanghai Skin Disease Hospital, School of Medicine, Tongji University

IPD SHARING:
Plan to Share IPD: Undecided